CLINICAL TRIAL: NCT01427309
Title: Efficacy Study of Fluzone® High-Dose Vaccine Compared With Fluzone® Vaccine In Elderly Adults
Brief Title: A Study of Fluzone® High-Dose Vaccine Compared With Fluzone® Vaccine In Elderly Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIM12; U1111-1120-1300 (Other: WHO)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Influenza; Trivalent Inactivated Influenza Vaccine; High-Dose Trivalent Inactivated Influenza Vaccine; Fluzone® High-Dose; Influenza vaccines
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose Trivalent Inactivated Influenza Vaccine (Experimental): Participants will receive an injection of High Dose Trivalent Inactivated Influenza Vaccine
  Interventions: Biological: High Dose Trivalent Inactivated Influenza Vaccine
- Trivalent Inactivated Influenza Vaccine (Active Comparator): Participants will receive an injection of the Trivalent Inactivated Influenza vaccine
  Interventions: Biological: Trivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: High Dose Trivalent Inactivated Influenza Vaccine — 0.5 mL Intramuscular
  Other Names: Fluzone® High Dose
  Arms: High Dose Trivalent Inactivated Influenza Vaccine
Biological: Trivalent Inactivated Influenza Vaccine — 0.5 mL, Intramuscular
  Other Names: Fluzone®
  Arms: Trivalent Inactivated Influenza Vaccine

SUMMARY:
The aim of this study is to determine the efficacy of Fluzone High-Dose compared to standard dose Fluzone for laboratory-confirmed or culture-confirmed influenza caused by influenza types/subtypes that are similar (for laboratory-confirmed) or antigenically similar (for culture-confirmed) to those contained in the respective annual vaccine formulations.

Primary Objective:

* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to laboratory-confirmed influenza caused by any influenza viral types/subtypes, associated with the occurrence of a protocol-defined influenza-like-illnesses (ILI).

Secondary Objectives:

* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to laboratory-confirmed influenza, caused by any influenza viral types/subtypes, associated with the occurrence of a protocol-defined ILI.
* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to culture-confirmed influenza, caused by any influenza viral types/subtypes, associated with the occurrence of a protocol-defined ILI.
* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to culture-confirmed influenza caused by viral types/subtypes antigenically similar to those contained in the respective annual vaccine formulations, associated with the occurrence of a modified Centers for Disease Control and Prevention (CDC)-defined ILI.
* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to culture-confirmed influenza caused by any influenza viral types/subtypes, associated with the occurrence of a modified CDC-defined ILI.
* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to culture-confirmed influenza caused by viral types/subtypes antigenically similar to those contained in the respective annual vaccine formulations, associated with the occurrence of a respiratory illness.
* To compare the clinical efficacy of Fluzone High-Dose to that of Fluzone in elderly adults, with respect to culture-confirmed influenza caused by any influenza viral types/subtypes, associated with the occurrence of a respiratory illness.

DETAILED DESCRIPTION:
The trial will span 2 influenza seasons. Each study year, participants will be randomized to receive one dose of either Fluzone® High-Dose or Fluzone® vaccine prior to the start of the influenza season and will be followed until the end of each season.

The duration of each participant's participation in the respective study year will be 6 to 8 months, depending on the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years on the day of vaccination
* Informed consent form signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination), or planned participation during each year of the trial period, in another clinical trial investigating a vaccine, drug, medical device, or medical procedure (Note: Concomitant participation in an observational trial is acceptable)
* Vaccination against influenza in the 6 months preceding the trial vaccination
* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone High-Dose or Fluzone vaccine or to a vaccine containing any of the same substances
* Personal history of Guillain-Barré Syndrome
* Dementia or any other cognitive condition at a stage that could interfere with following the trial procedures
* Thrombocytopenia contraindicating intramuscular (IM) vaccination, as judged by the investigator
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination, as judged by the investigator
* Current alcohol abuse or drug addiction
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Moderate or severe acute illness with or without fever (oral temperature > 99.0ºF [> 37.2ºC]). If this contraindication exists, vaccination will be deferred until the individual has been medically stable and/or afebrile (temperature ≤ 99.0 ºF [≤ 37.2ºC]) for at least 24 hours
* Signs and symptoms of an acute infectious respiratory illness. If this exists, vaccination will be deferred until the symptoms resolve.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31989 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (99):
- United States (91):
  - Mobile, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Harrisburg, Arkansas
  - Anaheim, California
  - La Mesa, California
  - Oceanside, California
  - Redding, California
  - San Diego, California
  - Santa Rosa, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Milford, Connecticut
  - Brooksville, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Crystal River, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Pembroke Pine, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - Stockbridge, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Lenexa, Kansas
  - Newton, Kansas
  - Overland Park, Kansas
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Lexington, Kentucky
  - Columbia, Maryland
  - Elkridge, Maryland
  - Rockville, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - Edina, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Bellevue, Nebraska
  - Omaha, Nebraska
  - Las Vega, Nevada
  - Newington, New Hampshire
  - Edison, New Jersey
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Endwell, New York
  - Rochester, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Idaho Falls, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Norman, Oklahoma
  - Erie, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scranton, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Clinton, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Bristol, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Salt Lake City, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Norfolk, Virginia
  - Williamsburg, Virginia
  - Winchester, Virginia
- Canada (6):
  - Coquitlam, British Columbia
  - Mount Pearl, Newfoundland and Labrador
  - Truro, Nova Scotia
  - Greater Sudbury, Ontario
  - Toronto, Ontario
  - Sherbrooke, Quebec
- Puerto Rico (2):
  - Bayamón
  - San Juan

REFERENCES:
- [Result] DiazGranados CA, Dunning AJ, Kimmel M, Kirby D, Treanor J, Collins A, Pollak R, Christoff J, Earl J, Landolfi V, Martin E, Gurunathan S, Nathan R, Greenberg DP, Tornieporth NG, Decker MD, Talbot HK. Efficacy of high-dose versus standard-dose influenza vaccine in older adults. N Engl J Med. 2014 Aug 14;371(7):635-45. doi: 10.1056/NEJMoa1315727. PMID 25119609
- [Derived] Becker DL, Chit A, DiazGranados CA, Maschio M, Yau E, Drummond M. High-dose inactivated influenza vaccine is associated with cost savings and better outcomes compared to standard-dose inactivated influenza vaccine in Canadian seniors. Hum Vaccin Immunother. 2016 Dec;12(12):3036-3042. doi: 10.1080/21645515.2016.1215395. Epub 2016 Sep 26. PMID 27669017
- [Derived] Dunning AJ, DiazGranados CA, Voloshen T, Hu B, Landolfi VA, Talbot HK. Correlates of Protection against Influenza in the Elderly: Results from an Influenza Vaccine Efficacy Trial. Clin Vaccine Immunol. 2016 Jan 13;23(3):228-35. doi: 10.1128/CVI.00604-15. PMID 26762363
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 06 September through 09 October 2011 for Year 1; and 09 through 21 October 2012 for Year 2 at 126 sites in the United States and Canada.
Pre-assignment Details: A total of 31,989 participants were enrolled 31,983 were randomized and vaccinated in this study.
Groups:
- Fluzone® High Dose Vaccine (Year 1); Fluzone® High Dose Vaccine (Year 2): Adults ≥65 years of age received one dose of Fluzone High Dose vaccine
- Fluzone® Vaccine (Year 1); Fluzone® Vaccine (Year 2): Adults ≥65 years of age received one dose of Fluzone vaccine
Period: Overall Study
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Started | 7253 | 7244 | 8737 | 8749
Completed | 6881 | 6837 | 8376 | 8373
Not Completed | 372 | 407 | 361 | 376
Not completed — Lost to Follow-up | 130 | 145 | 122 | 135
Not completed — Protocol Violation | 42 | 69 | 125 | 124
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Serious adverse event | 52 | 45 | 50 | 61
Not completed — Withdrawal by Subject | 148 | 148 | 61 | 55

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) as randomized, groups the participants according to the vaccine they were randomized to receive in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2) | Total
Number analyzed (Participants) | 7253 | 7244 | 8737 | 8749 | 31983
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 7253 | 7244 | 8737 | 8749 | 31983
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (5.88) | 73.2 (5.82) | 73.3 (5.74) | 73.4 (5.85) | 73.3 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4085 | 4041 | 5046 | 4922 | 18094
  Male | 3168 | 3203 | 3691 | 3827 | 13889
Region of Enrollment [Number; unit: Participants]
  United States | 6953 | 6944 | 8315 | 8326 | 30538
  Canada | 300 | 300 | 422 | 423 | 1445

OUTCOME MEASURES:

1. Primary Outcome: Occurrences of Culture- or Polymerase Chain Reaction (PCR)-Confirmed Influenza Caused by Any Influenza Viral Types/Subtypes, in Association With a Protocol-defined Influenza-like Illness (ILI).
Description: Influenza positive cultures were confirmed using direct immunofluorescence techniques with influenza type-specific antibodies. 3 culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney cells, Classic Flu A and B culture using Rhesus Monkey Kidney cells, and R Mix Flu A and B culture). The initial molecular test (PCR) was the validated ProFlu+™ assay by Prodesse, Inc., Waukesha, WI, which had been approved by the Food and Drug Administration through a 510K evaluation for specific detection of Influenza A, B or Respiratory Syncytial Virus.
  A protocol-defined influenza-like illness was determined by the occurrence of at least 1 of the following respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing; concurrently with at least one of the following systemic symptoms: fever (defined as temperature > 99.0°F [> 37.2°C]), chills (shivering), tiredness (fatigue), headache, or myalgia (muscle aches).
Time Frame: ≥14 days post-vaccination
Population: Clinical efficacy was assessed in subjects who met all eligibility criteria, received the vaccine they were randomized to, had successful surveillance contact, did not received additional influenza vaccinations and did not have protocol deviations likely to impact their responses for the primary and secondary endpoints (Per-protocol analysis set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 23 | 42 [0 to 0] | 204 [0 to 0] | 258 [0 to 0]

2. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Influenza Viral Types/Subtypes That Are Antigenically Similar to Those Contained in the Vaccine Formulations, in Association With a Protocol-defined Influenza-like Illness (ILI)
Description: Influenza positive cultures were confirmed by using direct immunofluorescence techniques with influenza type-specific (i.e., for Influenza A and Influenza B) antibodies. For culture confirmation of influenza, 3 different culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney [MDCK] cells, Classic Flu A and B culture using Rhesus Monkey Kidney [RhMK] cells, and R Mix Flu A and B culture. For antigenic similarity determinations, a standard hemagglutination inhibition test using a panel of ferret antisera (ferret antigenicity testing) was used.
Time Frame: ≥14 days post-vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 2 | 7 [0 to 0] | 61 [0 to 0] | 85 [0 to 0]

3. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Any Influenza Viral Types/Subtypes, in Association With a Protocol-defined Influenza-like Illness
Description: For culture confirmation of influenza, 3 different culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney [MDCK] cells, Classic Flu A and B culture using Rhesus Monkey Kidney [RhMK] cells, and R Mix Flu A and B culture).
  A protocol-defined influenza-like illness (ILI) was determined by the occurrence of at least one of the following respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing; concurrently with at least one of the following systemic symptoms: fever (defined as temperature > 99.0°F [> 37.2°C]), chills (shivering), tiredness (fatigue), headache, or myalgia (muscle aches).
Time Frame: ≥14 days post-vaccination
Population: Occurrences of culture-confirmed influenza caused by any influenza viral types/subtypes, in association with a protocol-defined influenza-like illness was assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 20 | 33 [0 to 0] | 185 [0 to 0] | 234 [0 to 0]

4. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Influenza Viral Types/Subtypes That Are Antigenically Similar to Those Contained in the Vaccine Formulations, in Association With a Modified CDC-defined Influenza-like Illness.
Description: Influenza positive cultures were confirmed by using direct immunofluorescence techniques with influenza type-specific antibodies. For culture confirmation of influenza, 3 different culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney cells, Classic Flu A and B culture using Rhesus Monkey Kidney cells, and R Mix Flu A and B culture). For antigenic similarity determinations, a standard hemagglutination inhibition test using a panel of ferret antisera (ferret antigenicity testing) was used.
  The modified Centers for Disease Control and Prevention-defined influenza-like illness is the occurrence of fever (defined as temperature > 99.0°F [> 37.2°C]) with cough or sore throat.
Time Frame: ≥14 days post-vaccination
Population: Occurrences of culture-confirmed influenza caused by influenza viral types/subtypes that are antigenically similar to those contained in the vaccine formulations, in association with a modified CDC-defined influenza-like illness were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 0 | 3 [0 to 0] | 22 [0 to 0] | 42 [0 to 0]

5. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Any Influenza Viral Types/Subtypes, in Association With a Modified CDC-defined Influenza-like Illness
Description: as for outcome 4
Time Frame: ≥14 days post-vaccination
Population: Occurrences of culture-confirmed influenza caused by any influenza viral types/subtypes, in association with a modified CDC-defined influenza-like illness were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 7 | 7 [0 to 0] | 77 [0 to 0] | 103 [0 to 0]

6. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Influenza Viral Types/Subtypes That Are Antigenically Similar to Those Contained in the Vaccine Formulations, in Association With a Respiratory Illness
Description: Influenza positive cultures were confirmed by using direct immunofluorescence techniques with influenza type-specific antibodies. For culture confirmation of influenza, 3 different culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney cells, Classic Flu A and B culture using Rhesus Monkey Kidney cells, and R Mix Flu A and B culture). For antigenic similarity determinations, a standard hemagglutination inhibition test using a panel of ferret antisera (ferret antigenicity testing) was used.
  Respiratory illness was defined as the occurrence of a new onset (or exacerbation of a pre-existing condition/symptom) of one or more of the following symptoms (that persist for or reoccur after a period of at least 12 hours): sneezing, stuffy or runny nose (nasal congestion), sore throat, cough, sputum production, wheezing, or difficulty breathing.
Time Frame: ≥14 days post-vaccination
Population: Occurrences of culture-confirmed influenza caused by influenza viral types/subtypes that are antigenically similar to those contained in the vaccine formulations, in association with a respiratory illness were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 7 | 9 [0 to 0] | 78 [0 to 0] | 109 [0 to 0]

7. Secondary Outcome: Occurrences of Culture-confirmed Influenza Caused by Any Influenza Viral Types/Subtypes, in Association With a Respiratory Illness
Description: Influenza positive cultures were confirmed by using direct immunofluorescence techniques with influenza type-specific (i.e., for Influenza A and Influenza B) antibodies. For culture confirmation of influenza, 3 different culture methods were utilized for each NP sample (Classic Flu A and B culture using Madin Darby Canine Kidney cells, Classic Flu A and B culture using Rhesus Monkey Kidney cells, and R Mix Flu A and B culture).
  Respiratory illness is defined as the occurrence of a new onset (or exacerbation of a pre-existing condition/symptom) of one or more of the following symptoms (that persist for or reoccur after a period of at least 12 hours): sneezing, stuffy or runny nose (nasal congestion), sore throat, cough, sputum production, wheezing, or difficulty breathing.
Time Frame: ≥14 days post-vaccination
Population: Occurrences of culture-confirmed influenza caused by any influenza viral types/subtypes, in association with a respiratory illness were assessed in the Per-Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7209 | 7207 | 8683 | 8704
Participants | 38 | 44 [0 to 0] | 238 [0 to 0] | 294 [0 to 0]

8. Other Pre Specified Outcome: Safety Overview After Injection With Either Fluzone High Dose or Fluzone Vaccine Through the End of Surveillance Period
Description: All serious adverse events, including deaths and adverse events (AEs) of special interest (Guillain Barre Syndrome, Bell's Palsy, encephalitis/myelitis, optic neuritis, Stevens Johnson Syndrome, and toxic epidermal necrolysis) were collected.
Time Frame: Day 0 up to Day 240 post-vaccination
Population: Safety was assessed in the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Number analyzed (Participants) | 7254 | 7243 | 8738 | 8748
Participants
  Serious adverse events (SAE) | 680 | 704 [0 to 0] | 643 [0 to 0] | 738 [0 to 0]
  Death | 48 | 40 [0 to 0] | 35 [0 to 0] | 44 [0 to 0]
  Adverse events of special interest | 2 | 2 [0 to 0] | 1 [0 to 0] | 4 [0 to 0]
  Guillain Barré Syndrome | 0 | 0 [0 to 0] | 0 [0 to 0] | 1 [0 to 0]
  Bell's palsy | 0 | 2 [0 to 0] | 1 [0 to 0] | 3 [0 to 0]
  Encephalitis/myelitis | 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Optic neuritis | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Stevens Johnson syndrome | 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Toxic epidermal necrolysis | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  SAE leading to study discontinuation | 52 | 45 [0 to 0] | 47 [0 to 0] | 58 [0 to 0]
  Related SAE | 1 | 0 [0 to 0] | 2 [0 to 0] | 0 [0 to 0]
  Related SAE leading to study discontinuation | 0 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: All serious adverse events, including deaths and adverse events (AEs) of special interest were collected from Day 0 (post-vaccination) up to Day 240 post-vaccination.
Description: The total number (N) data for the serious adverse events were presented for each study year according to the study vaccine actually recieved by the participants - the Full (as treated) Analysis Set.
Arm/Group | Fluzone® High Dose Vaccine (Year 1) | Fluzone® Vaccine (Year 1) | Fluzone® High Dose Vaccine (Year 2) | Fluzone® Vaccine (Year 2)
Serious Adverse Events (participants affected / at risk) | 680/7254 | 704/7243 | 643/8738 | 738/8748
Other Adverse Events (participants affected / at risk) | 0/7254 | 0/7243 | 0/8738 | 0/8748
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone® High Dose Vaccine (Year 1) (N=7254) | Fluzone® Vaccine (Year 1) (N=7243) | Fluzone® High Dose Vaccine (Year 2) (N=8738) | Fluzone® Vaccine (Year 2) (N=8748)
Anaemia (Blood and lymphatic system disorders) | 8 | 4 | 9 | 7
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 4 | 1 | 3 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 7 | 11 | 9
Angina pectoris (Cardiac disorders) | 2 | 8 | 5 | 5
Angina unstable (Cardiac disorders) | 2 | 9 | 8 | 5
Aortic valve disease mixed (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 2
Arrhythmia (Cardiac disorders) | 4 | 2 | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 28 | 29 | 23 | 38
Atrial flutter (Cardiac disorders) | 3 | 2 | 4 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 2 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1 | 2
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 5 | 4 | 2 | 2
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 6 | 1 | 0 | 5
Cardiac disorder (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 2 | 4
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 15 | 22 | 19 | 29
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 1 | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 2 | 3
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 14 | 18 | 16 | 18
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 4 | 2 | 3 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 2 | 2
Heart valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 2
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 21 | 21 | 14 | 10
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 2
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 3 | 4
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 3 | 1 | 3
Tachycardia (Cardiac disorders) | 2 | 1 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 2 | 1 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 5 | 2 | 7
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 6 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 2 | 2 | 3 | 4
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Colonic stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 5 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Gastritis (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 7 | 5 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Lumbar hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 5 | 2 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 2 | 0 | 5
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 5 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 10 | 4 | 3
Spigelian hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 1 | 2
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 2
Chest discomfort (General disorders) | 1 | 2 | 1 | 2
Chest pain (General disorders) | 42 | 27 | 18 | 16
Death (General disorders) | 0 | 3 | 0 | 2
Device dislocation (General disorders) | 0 | 0 | 0 | 2
Device failure (General disorders) | 0 | 0 | 0 | 1
Device lead damage (General disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 2 | 1 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Genaralized oedema (General disorders) | 0 | 0 | 1 | 0
Hernia (General disorders) | 1 | 0 | 0 | 1
Hernia obstructive (General disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Implant site inflammation (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 1 | 0
Ischaemic ulcer (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 6 | 3 | 2 | 4
Oedema peripheral (General disorders) | 2 | 1 | 1 | 1
Pelvic mass (General disorders) | 0 | 0 | 0 | 1
Pneumatosis (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0
Surgical failure (General disorders) | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 8 | 3
Cholecystitis acute (Hepatobiliary disorders) | 3 | 2 | 3 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 7 | 5 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 4 | 3 | 4
Arthritis bacterial (Infections and infestations) | 1 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 1 | 0
Atypical myocobacterial pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 5 | 4 | 9 | 5
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 12 | 9 | 8 | 12
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 3 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 1 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1 | 1
Diabetic gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 8 | 5 | 5 | 11
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 1
Enterocolitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastric ulcer helicobacter (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 6 | 5 | 9
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 2 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 3 | 6
Kidney infection (Infections and infestations) | 0 | 1 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 2 | 6
Localised infection (Infections and infestations) | 2 | 2 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 1
Peridiverticular abscess (Infections and infestations) | 0 | 0 | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 28 | 44 | 35 | 44
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 2
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 2
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 2
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 2 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 3 | 0 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 4 | 3 | 5 | 5
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 3
Tracheobronchitis (Infections and infestations) | 2 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 8 | 5 | 16
Urosepsis (Infections and infestations) | 5 | 3 | 0 | 4
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 4
Viral labyrinthitis (Infections and infestations) | 0 | 0 | 2 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 5 | 5 | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Ear injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 5 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 6 | 5 | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 8 | 4 | 5 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 2 | 4 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2
Injury (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 3
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 3 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 4 | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 5
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 2
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 | 7 | 7 | 4
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 48 | 29 | 50 | 35
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 0 | 3
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 11 | 7 | 7
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 4 | 5
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastrinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Laryngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung carcinoma cell type unspecified stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 11 | 6 | 3
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myeloma recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2 | 3 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 2
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 2 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 2 | 4 | 0
Cerebral amyloid angiopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1 | 2 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1 | 0 | 2
Cerebral Ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 20 | 19 | 13 | 21
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 3 | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 1 | 2 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 2 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 3 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 3 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 3 | 3 | 2
Radiculopathy (Nervous system disorders) | 1 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 4 | 1 | 1
Syncope (Nervous system disorders) | 18 | 19 | 15 | 16
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Transient global amnesia (Nervous system disorders) | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 12 | 15 | 9 | 12
VIIth nerve paralysis (Nervous system disorders) | 0 | 2 | 1 | 3
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 1 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 2 | 5 | 4
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Bladder fibrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 2 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 2 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 5 | 2 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 1 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 1 | 1 | 4
Renal failure acute (Renal and urinary disorders) | 8 | 5 | 11 | 14
Renal failure chronic (Renal and urinary disorders) | 4 | 2 | 1 | 3
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 3 | 2 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Genital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 6 | 7
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 5
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 21 | 13 | 15 | 36
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 6 | 13
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Activities of daily living impaired (Social circumstances) | 1 | 0 | 0 | 0
Colostomy (Surgical and medical procedures) | 1 | 0 | 0 | 1
Face lift (Surgical and medical procedures) | 0 | 1 | 0 | 0
Implantable defibrillator removal (Surgical and medical procedures) | 1 | 0 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 0 | 0 | 1
Renal surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0 | 2
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 5 | 3 | 5 | 6
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 2 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 2 | 0
Aortic rupture (Vascular disorders) | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 2 | 2 | 2 | 2
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Arterial stenosis limb (Vascular disorders) | 1 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 1 | 0 | 3
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 5 | 1 | 6
Embolism venous (Vascular disorders) | 0 | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 4 | 2 | 1 | 0
Hypertension (Vascular disorders) | 8 | 4 | 4 | 3
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 8 | 4 | 2 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Infarction (Vascular disorders) | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 1 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 5 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 2 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 3 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 1 | 2
Shock (Vascular disorders) | 0 | 0 | 1 | 0
Steal syndrome (Vascular disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No